CLINICAL TRIAL: NCT03204760
Title: Steroids In The Management Of Acute Asthma Exacerbations In Children, Which Form Is More Suitable?
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Eman Alfy Ellia, Resident pediatrician , Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eman Alfy Ellia
Record Dates: First submitted 2017-06-22; First posted 2017-07-02 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Steroids In Management Of Acute Asthma Exacerbations
MeSH Terms: interventions — Dexamethasone; Solutions; Injections; Prednisolone

STUDY DESIGN:
Intervention Model Description: Children with mild to moderate asthma exacerbation will be given the first dose of salbutamol and will be reassessed after 20 min by the emergency department attending. If further salbutamol is needed, subjects automatically will receive the second dose 20 min apart and receive either single dose of intramuscular dexamethasone (0.6 mg/kg to a maximum of 18 mg) or prednisolone for 3 days (1 mg/kg to a maximum of 40 mg), given orally in two devided doses .
  A repeat physical examination will be performed, including oxygen saturation, vital signs, PRAM, PEFR after the 3rd dose of salbutamol and at the end of the third day to evaluate the effect of prednisolone and dexamethasone on the improvement of asthma scores. Patient compliance to prednisolone therapy for three days will be also recorded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexamethasone (Experimental): Dexamethasone is a long-acting glucocorticoid with a half-life of 36 to 72 hours . It has been used safely in children with croup and bacterial meningitis . It is well absorbed both orally and parenterally .Single dose of intramuscular dexamethasone (0.6 mg/kg to a maximum of 18 mg).
  Interventions: Drug: Dexamethasone 8Mg Solution for Injection
- prednisolone (Experimental): Prednisolone is relatively short acting with a half-life of 12 to 36 hours, thereby requiring daily dosing. Outpatient steroid therapy is effective once compliance is assured.. Prolonged treatment course, vomiting, and a bitter taste may reduce patient compliance with prednisolone. Oral prednisolone for 3 days (1 mg/kg to a maximum of 40 mg), given orally in two devided doses .
  Interventions: Drug: Prednisolone Oral, Per 5 Mg

INTERVENTIONS:
Drug: Dexamethasone 8Mg Solution for Injection — Effect single dose of intramuscular dexamethasone (0.6 mg/kg to a maximum of 18 mg) in the treatment of mild to moderate acute asthma exacerbations in children
  Arms: dexamethasone
Drug: Prednisolone Oral, Per 5 Mg — Effect of prednisolone for 3 days (1 mg/kg to a maximum of 40 mg), given orally in two devided doses in the treatment of mild to moderate acute asthma exacerbations in children.
  Arms: prednisolone

SUMMARY:
The aim of this study is to compare the efficacy of a single dose of intramuscular dexamethasone versus 3 days of twice-daily oral prednisolone in the management of mild to moderate asthma exacerbations in children and test whether this single dose of intramuscular dexamethasone 0.6 mg/kg (max. 18 mg) is equal to prednisolone 1 mg/kg/day (max. 40 mg) in the treatment of exacerbations of asthma in children, as measured by the Pediatric Respiratory Assessment Measure (PRAM).

DETAILED DESCRIPTION:
This study will be performed in Assiut university Children Hospital and will include patients with asthma exacerbations presented to the emergency department for three months. All children presenting to the emergency department with mild to moderate asthma exacerbations will be assessed to decide if the child needs treatment with salbutamol. Before starting treatment the Pediatric Respiratory Assessment Measure (PRAM), vital signs, and oxygen saturation will be recorded. Peak expiratory flow rate (PEFR) will also be recorded if the patient was 6 years or older.

Children with mild to moderate asthma exacerbation will be given the first dose of salbutamol and will be reassessed after 20 min by the emergency department attending. If further salbutamol is needed, subjects automatically will receive the second dose 20 min apart and receive either single dose of intramuscular dexamethasone (0.6 mg/kg to a maximum of 18 mg) or oral prednisolone for 3 days (1 mg/kg to a maximum of 40 mg), given orally .

A repeat physical examination will be performed, including oxygen saturation, vital signs, PRAM, PEFR after the 3rd dose of salbutamol and at the end of the third day to evaluate the effect of prednisolone and dexamethasone on the improvement of asthma scores. Patient compliance to prednisolone therapy for three days will be also recorded.

This study will be performed in Pediatric hospital - Assiut university and will include patients with asthma exacerbations presented to the emergency department for three months.

ELIGIBILITY:
Inclusion Criteria:

* Ages 2 to 16 years
* Background history of asthma
* Presentation with an asthma exacerbation requiring repeated salbutamol after 20 minutes.

Exclusion Criteria:

* Less than 2 years old or over 16 years
* Critical or life-threatening asthma
* Known tuberculosis exposure
* Active varicella or herpes simplex infection
* Documented concurrent infection with Respiratory syncytial virus
* Fever >39.5°C
* Use of oral corticosteroids in the previous four weeks
* Concurrent stridor
* Significant co-morbid disease: lung, cardiac, immune, liver, endocrine, neurological or psychiatric

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2018-02-28 (Estimated)

PRIMARY OUTCOMES:
The Pediatric Respiratory Assessment Measure (PRAM) | PRAM score is assessed at the end of the third day to evaluate the effect of prednisolone and dexamethasone on the improvement of asthma scores.
  The Pediatric Respiratory Assessment Measure (PRAM) , a validated, responsive and reliable tool to determine asthma severity in children aged 2 to 16 years, appears to be the most appropriate as an application in the emergency care setting .
  The PRAM score consists of five components and has a maximum total of 12 points: suprasternal retractions (0 to 2), scalene muscle contraction (0 to 2), air entry (0 to 3), wheezing (0 to 3) and O2 saturation (0 to 2) .

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa M. El-Saied, Ph.D.of pediatrics, Study Chair — Assiut University -Faculty of medecin( Pediaric department)
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No